CLINICAL TRIAL: NCT04373746
Title: Accuracy of the NICCI™ Monitor in Providing Beat-to-beat Non-invasive Blood Pressure Readings in Children and Adolescents
Brief Title: Accuracy of the NICCI™ Monitor in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000959
Record Dates: First submitted 2020-04-22; First posted 2020-05-04 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Surgery; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 10-40 kg (Experimental): Patients undergoing major surgery that weigh between 10-20 kg.
  Interventions: Device: NICCI
- 40-80 kg (Experimental): Patients undergoing major surgery that weigh between 40-80 kg.
  Interventions: Device: NICCI

INTERVENTIONS:
Device: NICCI — Non-invasive beat-to-beat blood pressure monitor capable of producing a waveform similar to an invasive arterial line.

SUMMARY:
This is a prospective study that will compare the blood pressure readings from an arterial cannula with those obtained non-invasively by the NICCI device. The study will enroll 50 patients into each of three weight ranges: 10-20 kg, 20-40 kg, and 40-80 kg.

The NICCI, Pulsion/GETINGE uses novel technology to provide a continuous estimation of BP displayed as a waveform similar to that seen with an invasive arterial cannula, but is totally non-invasive by using the fingers. The patient rests their hand on the device, which is about the size of a computer mouse, and then a blood pressure cuff goes around their upper arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring anesthetic care and in whom an indwelling arterial cannula will be placed for the surgical procedure.

Exclusion Criteria:

* Patients with history of a peripheral neurologic or neuropathic disorder
* Patients in whom the upper extremity cannot be used for blood pressure monitoring
* Patients in whom an invasive arterial cannula cannot be placed
* Patients with vascular implants at the sites of non-invasive blood pressure measurement (fingers and upper arm of the examined arm)
* Edematous patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 10-40 kg: Patients undergoing major surgery that weigh between 10-40 kg.
  NICCI: Non-invasive beat-to-beat blood pressure monitor capable of producing a waveform similar to an invasive arterial line.
Period: Overall Study
Arm/Group | 10-40 kg | 40-80 kg
Started | 31 | 51
Completed | 24 | 44
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10-40 kg | 40-80 kg | Total
Number analyzed (Participants) | 24 | 44 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 44 | 68
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 11 (4) | 15 (2) | 14 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 23 | 35
  Male | 12 | 21 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 6 | 6
  White | 23 | 35 | 58
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 44 | 68
Weight [Mean (Standard Deviation); unit: kilograms] | 30 (8) | 56 (10) | 48 (15)
Height [Mean (Standard Deviation); unit: centimeters] | 134 (19) | 162 (9) | 153 (19)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 17 (2) | 22 (4) | 20 (4)
Patient position [Count of Participants; unit: Participants]
  Prone | 18 | 40 | 58
  Supine | 6 | 3 | 9
  Lateral | 0 | 1 | 1
ASA physical class [Count of Participants; unit: Participants] — American Society of Anesthesiologists classification system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. ASA 1 = healthy patient, 2 = mild systemic disease, 3 = severe systemic disease, 4 = severe systemic disease that is a constant threat to life.
  Participants
    1 | 1 | 8 | 9
    2 | 10 | 22 | 32
    3 | 10 | 13 | 23
    4 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Difference in Blood Pressure
Description: The absolute difference of the SBP, DBP, and MAP values from the arterial cannula (AC) and NICCI device were calculated. Instead of the directional difference (positive or negative), the absolute difference was used to avoid affecting the data when calculating the mean and standard deviation (SD) of the differences. For instance, if the reading from the NICCI device was 5 mm Hg above or below the reading from the AC, a value of 5 mm Hg was used and not -5 mm Hg or +5 mm Hg.
Time Frame: 2-8 hours (average length of major surgery)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 10-40 kg | 40-80 kg
Number analyzed (Participants) | 24 | 44
mm Hg
  SBP | 11 (9) | 10 (8)
  DBP | 10 (7) | 9 (7)
  MAP | 10 (7) | 9 (7)

2. Secondary Outcome: Percentage of BP Values From the NICCI Device That Were ≤ 5 mm Hg the Values Obtained From the AC
Description: The absolute difference of the SBP, DBP, and MAP values from the arterial cannula (AC) and NICCI device were calculated. Instead of the directional difference (positive or negative), the absolute difference was used to avoid affecting the data when calculating the mean and standard deviation (SD) of the differences. For instance, if the reading from the NICCI device was 5 mm Hg above or below the reading from the AC, a value of 5 mm Hg was used and not -5 mm Hg or +5 mm Hg. We also calculated the percentage of BP values from the NICCI device that were ≤ 5 mm Hg, ≤ 10 mm Hg, and > 10 mm Hg from the values obtained from the AC.
Time Frame: 2-8 hours (average length of major surgery)
Population: The study team analyzed pairs of SBP, DBP, and MAP values from the NICCI device and the arterial canula.
Measure: Number; unit: percentage of NICCI readings
Units Other Than Participants: pairs of SBP, DBP, and MAP values
Arm/Group | 10-40 kg | 40-80 kg
Number analyzed (Participants) | 24 | 44
Number analyzed (pairs of SBP, DBP, and MAP values) | 146562 | 383126
percentage of NICCI readings
  SBP | 32 | 35
  DBP | 35 | 39
  MAP | 31 | 31

3. Secondary Outcome: Percentage of BP Values From the NICCI Device That Were ≤ 10 mm Hg the Values Obtained From the AC
Description: as for outcome 2
Time Frame: 2-8 hours (average length of major surgery)
Population: The study team analyzed pairs of SBP, DBP, and MAP values from the NICCI device and the arterial canula.
Measure: Number; unit: percentage of NICCI readings
Units Other Than Participants: pairs of SBP, DBP, and MAP values
Arm/Group | 10-40 kg | 40-80 kg
Number analyzed (Participants) | 24 | 44
Number analyzed (pairs of SBP, DBP, and MAP values) | 146562 | 383126
percentage of NICCI readings
  SBP | 57 | 60
  DBP | 60 | 67
  MAP | 56 | 56

4. Secondary Outcome: Percentage of BP Values From the NICCI Device That Were > 10 mm Hg From the Values Obtained From the AC
Description: as for outcome 2
Time Frame: 2-8 hours (average length of major surgery)
Population: The study team analyzed pairs of SBP, DBP, and MAP values from the NICCI device and the arterial canula.
Measure: Number; unit: percentage of NICCI readings
Units Other Than Participants: pairs of SBP, DBP, and MAP values
Arm/Group | 10-40 kg | 40-80 kg
Number analyzed (Participants) | 24 | 44
Number analyzed (pairs of SBP, DBP, and MAP values) | 146562 | 383126
percentage of NICCI readings
  SBP | 43 | 40
  DBP | 40 | 33
  MAP | 44 | 44

ADVERSE EVENTS:
Time Frame: 1 week after surgery
Arm/Group | 10-40 kg | 40-80 kg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/44
Other Adverse Events (participants affected / at risk) | 0/24 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT04373746/Prot_SAP_000.pdf